CLINICAL TRIAL: NCT07003425
Title: A Long-term Extension Study to Evaluate the Safety and Efficacy of APG777 in Patients With Atopic Dermatitis Previously Treated With APG777
Brief Title: A Long-term Safety and Efficacy Study Evaluating APG777 in Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Apogee Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APG777-202
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; APG777; Safety; Efficacy
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- APG777 - Long Term Extension Treatment - 12 Weeks (Experimental): Participants who achieve EASI 75 or a vIGA-AD (0, 1) at the end of the Parent Study Treatment Period, and who did not use topical rescue medication during the Parent Study will maintain the same dose regimen (dose and frequency of injections) from the Maintenance Period of the Parent Study (APG777-201).
  Interventions: Drug: APG777
- APG777 - Long Term Extension Treatment - 24 Weeks (Experimental): Participants who achieve EASI 75 or a vIGA-AD (0, 1) at the end of the Parent Study Treatment Period, and who did not use topical rescue medication during the Parent Study, will maintain the same dose regimen (dose and frequency of injections) from the Maintenance Period of the Parent Study (APG777-201).
  Interventions: Drug: APG777
- APG777 - Open Label Escape Arm (Experimental): Participants who do not achieve EASI 75 or a vIGA-AD (0, 1) at the end of the Parent Study Treatment Period, or who used topical rescue medication during the Parent Study, will be assigned to the open-label Escape Arm and will receive APG777 per protocol defined dosing regimen.
  Interventions: Drug: APG777

INTERVENTIONS:
Drug: APG777 — APG777 subcutaneous injection
  Arms: APG777 - Open Label Escape Arm
Drug: APG777 — APG777 subcutaneous injection every 12 weeks
  Arms: APG777 - Long Term Extension Treatment - 12 Weeks
Drug: APG777 — APG777 subcutaneous injection every 24 weeks
  Arms: APG777 - Long Term Extension Treatment - 24 Weeks

SUMMARY:
This is a multicenter, double-blind, Long-Term Extension (LTE) study to evaluate the long-term safety and efficacy of APG777 in patients with moderate-to-severe AD who have completed treatment in an APG777 Parent Study (NCT06395948).

The LTE study will consist of 3 periods: 1) Screening Visit will coincide with the last visit of the Maintenance Period in the Parent Study 2) Extended Treatment Period 3) Post-treatment Follow-up Period.

This study will be conducted in participants with atopic dermatitis (AD) who completed the Treatment Period in a prior APG777 study and who, in the opinion of the Investigator, would benefit from long-term treatment with APG777.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed the Treatment Period in a prior APG777 study and were, in the Investigator's opinion, compliant with the study protocol
* Participants who, in the Investigator's opinion, would benefit from long-term treatment with APG777
* Use the same non-prescription non-medicated emollient/moisturizer of their choice from the last day of the Parent Study and throughout the LTE study

Exclusion Criteria:

* Participants who have developed an AE while participating in the Parent Study. which, in the opinion of the Investigator or of the Medical Monitor, could indicate that continued treatment with APG777 may present an unreasonable risk for the patient
* Participants who terminated early from the Parent Study or permanently discontinued the study drug during the Parent Study
* Use of any of the prohibited medications in the Parent Study through Screening Visit (Visit 1) of the LTE study
* Presence of dermatologic conditions and/or comorbidities that might confound the diagnosis of AD and/or interfere with study assessments

Note: Additional protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events | Up to 3 years

SECONDARY OUTCOMES:
Percentage of Participants who achieve Eczema Area and Severity Index (EASI) 50, 75, 90, and 100 calculated based on Parent Study Baseline | Through Extended Treatment Period, an average of 2 years
Percentage of Participants who achieve a validated Investigator Global Assessment Atopic Dermatitis (vIGA AD) score of 0 (clear) or 1 (almost clear) and a ≥ 2-point reduction as calculated based on Parent Study Baseline. | Through Extended Treatment Period, an average of 2 years
Percentage of Participants who achieve ≥ 4-point improvement in the weekly mean of the daily Itch Numeric Rating Scale (I-NRS) as calculated based on Parent Study Baseline | Through Extended Treatment Period, an average of 2 years
Percentage of Participants who use Rescue Therapy | Through Extended Treatment Period, an average of 2 years
Percentage of Participants Who Continue to Exhibit EASI 75 | From Week 52 up to Through Extended Treatment Period, an average of 2 years
  Of the participants who achieve EASI 75 at Week 52 of the Parent Study, the percentage that continue to exhibit EASI 75 will be determined
Percentage of Participants Who Continue to Exhibit vIGA-AD Response | From Week 52 up to Through Extended Treatment Period, an average of 2 years
  Of the participants who achieve vIGA-AD of clear (0) or almost clear (1) and a ≥ 2-Point reduction at Week 52 of the Parent Study, the percentage that continue to exhibit the response will be determined.
Percentage of Participants Who Continue to Exhibit I-NRS Response | From Week 52 up to Through Extended Treatment Period, an average of 2 years
  Of the participants who achieve a ≥ 4 point improvement in the weekly mean of the daily I NRS at Week 52 of the Parent Study, the percentage that continue to exhibit the response will be determined.
Number of Participants who Discontinued Treatment Due to Treatment-Related TEAEs and SAEs | Up to 3 years
Serum Concentrations of APG777 Over Time | Up to 3 years
Predose Serum Concentrations of APG777 | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (35):
- United States (18):
  - Investigational Site, Fountain Valley, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, Coral Gables, Florida
  - Investigational Site, Margate, Florida
  - Investigational Site, Douglasville, Georgia
  - Investigational Site, Skokie, Illinois
  - Investigational Site, Bowling Green, Kentucky
  - Investigational Site, Detroit, Michigan
  - Investigational Site, Troy, Michigan
  - Investigational Site, New York, New York
  - Investigational Site, Wilmington, North Carolina
  - Investigational Site, Boardman, Ohio
  - Investigational Site, Mason, Ohio
  - Investigational Site, Portland, Oregon
  - Investigational Site, Nashville, Tennessee
  - Investigational Site, Dallas, Texas
  - Investigational Site, Frisco, Texas
  - Investigational Site, San Antonio, Texas
- Canada (9):
  - Investigational Site, Calgary, Alberta
  - Investigational Site, Edmonton, Alberta
  - Investigational Site, Fredericton, Brunswick
  - Investigational Site, Markham, Ontario
  - Investigational Site, Mississauga, Ontario
  - Investigational Site, Peterborough, Ontario
  - Investigational Site, Toronto, Ontario
  - Investigational Site, Montreal, Quebec
  - Investigational Site, Québec, Quebec
- Poland (8):
  - Investigational Site, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site, Lublin, Lublin Voivodeship
  - Investigational Site, Warsaw, Masovian Voivodeship
  - Investigational Site, Gdansk, Pomeranian Voivodeship
  - Investigational Site, Katowice, Silesian Voivodeship
  - Investigational Site, Sosnowiec, Silesian Voivodeship
  - Investigational Site, Krakow, Woj. Małopolskie
  - Investigational Site, Lodz